CLINICAL TRIAL: NCT03461952
Title: A Phase II Open Label, Randomized Non-Comparative Trial of Nivolumab Alone or in Combination With Ipilimumab for the Treatment of Patients With Advanced Hypermutated Solid Tumors Detected by a Blood Based Assay
Brief Title: Nivolumab Ipilimumab in Patients With hyperMutated Cancers Detected in Blood (NIMBLe)
Acronym: NIMBLe
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: cfDNA screening data found that the prevalence of POLE/POLD1 mutations was lower than expected. It was determined that there are no feasible options to amend this study in a fashion that would not be duplicative of other currently accruing trials.
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Cancer Research Institute, New York City (Other); Bristol-Myers Squibb (Industry); Personal Genome Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I235; 0001 (Other: Cancer Research Institute)
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab (Experimental): 240mg Q2W
  Interventions: Drug: Nivolumab
- Nivolumab + Ipilimumab (Experimental): Nivolumab 240mg Q2Wk + Ipilimumab 1mg/kg Q6W
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — 240mg
Drug: Ipilimumab — 1mg/kg
  Arms: Nivolumab + Ipilimumab

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of nivolumab alone or in combination with ipilimumab in patients with metastatic or unresectable tumors harbouring mutations in genes, POLE and POLD1. These mutations will be determined by plasma cfDNA. Nivolumab and ipilimumab have been given to patients across multiple types of cancer, and safe doses and schedules have been determined.

DETAILED DESCRIPTION:
Participants in this study have been diagnosed with metastatic or unresectable solid tumors that have a mutation in POLE and/or POLD1. Nivolumab alone or in conjunction with ipilimumab is predicted to be effective against tumors with POLE and/or POLD1 mutations as these genetic changes cause increased rates of mutations in the DNA of tumor cells. These high mutation rates have been associated with response to immunotherapy agents such as nivolumab and ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced (metastatic or unresectable) solid tumors.
* Patients must have received at least 1 standard cancer therapy for their tumor type and progressed on their most recent regimen; patients may be treatment naïve if they refuse standard treatment or there is no standard treatment for their cancer.
* Prior adjuvant/neoadjuvant therapy with curative intent is considered a prior therapy if disease recurrence occurs within at least 6 months.
* Patients may not have received prior immunotherapy
* Patients must consent to blood collection for testing after registration by a central reference laboratory.
* Patients must have clinically and/or radiologically documented disease with at least one lesion measurable as defined by RECIST 1.1.
* Patients must be ≥ 18 years of age.
* ECOG performance status 0 or 1.
* Patients must have adequate hematology and organ function
* Patient consent for screening must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Patients must have solid tumors that demonstrate POLE or POLD1 mutations identified at study entry via plasma cfDNA testing or tumor tissue testing for POLE and POLD1 mutations. A CLIA-certified testing of tumor tissue demonstrating POLE or POLD1 mutation can qualify for eligibility and randomization, however, plasma will be submitted for central cfDNA testing. In the event of discordance between tissue and central laboratory testing, the patient will continue in study but will not be included in the primary analysis. These patients will however be included in the secondary analysis.
* Patients must have recovered to ≤ grade 1 from all reversible toxicity related prior systemic or radiation therapy and have a 2 weeks washout.
* Previous major surgery is permitted provided that it has been at least 28 days prior to patient registration and that wound healing has occurred.
* White Blood Cells ≥ 2.0 x 109/L (2000/µL)
* Absolute neutrophils ≥ 1.5 x 109/L (1500/µL)
* Platelets ≥ 100 x 10^9/L (100 x103/µL)
* Hemoglobin ≥80 g/L* (8.0 g/dL)
* Bilirubin ≤ 1.5 x ULN (upper limit of normal)**
* AST and/or ALT ≤ 3 x ULN
* Serum creatinine ≤ 1.5 x ULN or: Creatinine clearance ≥40 mL/min
* Patients must be willing to consent to provision of archival tissue
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the trial.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient randomization.
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must have agreed to use a highly effective contraceptive method

Exclusion Criteria:

* Patients with a history of other untreated malignancies or malignancies, which required therapy within the past 2 years. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen may be eligible after consultation with the CCTG.
* Patients with primary CNS tumors are not eligible.
* Patients with active brain metastases or leptomeningeal metastases are not eligible. Patients with brain metastases are eligible if these have been treated and clinically stable. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents). Physiologic replacement doses of systemic corticoidsteroids are permitted, even if >10mg/day prednisone equivalents
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 14 days of study drug administration*
* Active or prior documented autoimmune or inflammatory disorders. Including, inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions considered to be of low risk for recurrence are permitted to enroll.
* History of hypersensitivity to nivolumab or ipilimumab or any excipient.
* Any previous treatment with a PD-1 or anti-PD-L1, anti-PD-L2 inhibitor, including nivolumab or an anti-CTLA4, including ipilimumab, or drug specifically targeting T-cell stimulation or immune checkpoint pathways.
* Patients with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol (including corticosteroid administration), or would put the patient at risk. This includes but is not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements.
  * Active infection requiring systemic therapy; (including any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) or tuberculosis or any infection requiring systemic therapy).
  * Active peptic ulcer disease or gastritis
  * Active pneumonitis.
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational anti-cancer agents.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects).
* Pregnant or lactating women.
* Men who are sexually active with women of childbearing potential and women of childbearing potential must agree to use adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, Study Chair — Thoracic Oncology and Immunotherapeutics, Columbia University Hospital
Locations (6):
- Columbia University Medical Center, New York, New York, United States
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 53 [31 to 75] | 53 [50 to 55] | 53 [31 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate by RECIST 1.1
Description: Objective Response Rate by RECIST 1.1: CR, PR, SD, or PD
Time Frame: 36 months
Population: The study was pre-maturely closed to accrual on August 2, 2019 following review of screening data which found that the prevalence of relavent mutations was lower than expected. Only 4 patients were accrued.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 2 | 2
Participants | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy. | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy.

2. Secondary Outcome: Efficacy as Measured by Objective Response Rate
Description: Will be reported using percentages over all randomized patients with 90% exact confidence intervals
Time Frame: 36 months
Population: The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 2 | 2
Participants | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy. | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy.

3. Secondary Outcome: Duration of Response
Description: Response rates will be reported using percentages over all patients who have received at least one dose of treatment with 90% exact CI of each arm in a non-comparative analysis
Time Frame: 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 2 | 2
Participants | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy. | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy.

4. Secondary Outcome: Number and Severity of Adverse Events Using CTCAE 5.0
Description: AE rates will be reported using percentages with 90% exact CI
Time Frame: 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 2 | 2
Participants | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy. | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy.

5. Secondary Outcome: Correlation Between POLE or POLD1 Mutations in Tumor and POLE or POLD1 Mutations in Blood
Description: Correlation between POLE or POLD1 mutations in tumor and POLE or POLD1 mutations in blood: Will be assessed by Fischer's exact test in each arm
Time Frame: 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 2 | 2
Participants | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy. | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy.

6. Secondary Outcome: To Evaluate Response by iRECIST
Description: iRECIST: iCR, iPR, iSD, iUPD, iUPD/PD
Time Frame: 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
Number analyzed (Participants) | 2 | 2
Participants | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy. | NA — The actual enrolment is extremely small for the study and any form of outcome measure will inevitability leak patients' privacy.

ADVERSE EVENTS:
Time Frame: 36 months.
Arm/Group | Nivolumab | Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=2) | Nivolumab + Ipilimumab (N=2)
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT03461952/Prot_SAP_001.pdf